CLINICAL TRIAL: NCT00106691
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Efficacy and Safety Study of Toremifene Citrate for the Prevention of Prostate Cancer in Men With High Grade Prostatic Intraepithelial Neoplasia (PIN)
Brief Title: Prostate Cancer Prevention Study for Men With High Grade PIN (Prostatic Intraepithelial Neoplasia)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: G300104
Record Dates: First submitted 2005-03-29; First posted 2005-03-30 (Estimated); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Preneoplastic Conditions; Prostatic Intraepithelial Neoplasia
Keywords: neoplasia; chemoprevention; cancer; premalignant; precancerous; Chemoprophylaxis; Intraepithelial Prostatic Neoplasia; Neoplasia, Prostatic Intraepithelial
MeSH Terms: conditions — Precancerous Conditions; Prostatic Intraepithelial Neoplasia; Neoplasms | interventions — Toremifene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20 mg Toremifene Citrate (Experimental): The subject takes one dose by mouth of the 20mg Toremifine Citrate tablet once a day for the length of the trial (360 days).
  Interventions: Drug: Toremifene 20 mg
- Placebo (Experimental): The subject takes a placebo tablet identical in appearance to the toremifene 20mg tablet, administered by mouth daily for 360 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Toremifene 20 mg — The subject takes one dose by mouth of the 20mg Toremifine Citrate tablet once a day for the length of the trial (360 days).
  Arms: 20 mg Toremifene Citrate
Drug: Placebo — The subject takes a placebo tablet identical in appearance to the toremifene 20mg tablet, administered by mouth daily for 360 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if toremifene citrate is effective and safe in the prevention of prostate cancer in men who have been diagnosed with high grade prostatic intraepithelial neoplasia (PIN).

DETAILED DESCRIPTION:
The purpose of this study is to determine if toremifene citrate is effective and safe in the prevention of prostate cancer in men who have been diagnosed with high grade prostatic intraepithelial neoplasia. Men who have ever been diagnosed with high grade PIN will be enrolled into an 36 month trial and will be assigned to either 20 mg of study drug or placebo per day. Subjects will undergo safety evaluations at Month 3, Month 6, Month 12, Month 18, Month 24, Month 30 and Month 36 along with prostate biopsies at Month 12 and Month 24 and Month 36 to determine efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary signed informed consent in accordance with institutional policies
* Be male, aged ≥ 30 years
* Have a diagnosis of high grade PIN from any previous prostate biopsy. The diagnosis of high grade PIN must be confirmed by the central pathologist
* Have had a prostate biopsy in the last 6 months with a minimum of 10 cores that shows no evidence of cancer as confirmed by the central pathologist; OR, have had 2 prostate biopsies (each with a minimum of 6 cores) in the 12 months prior to screening with at least one of the biopsies occurring within 6 months prior to the screening visit. Both biopsies should have no evidence of cancer as confirmed by the central pathologist
* Have a serum PSA of ≤ 10 ng/mL
* Agree to provide tablet containers for tablet counts and to complete a daily diary of study drug intake
* Agree to use an effective method of contraception, if the partner is of child-bearing age, while on study and for 30 days after the last dose of study medication
* Have adequate bone marrow, liver and renal function:

  * White Blood Cell (WBC) Count ≥ 3,000/mm3;
  * Platelet Count ≥ 100,000/mm3;
  * Bilirubin ≤ 1.5 mg/dL;
  * AST and ALT < 2x upper limit of normal;
  * Serum Creatinine ≤ 2.0 mg%

Exclusion Criteria:

* Previous exposure to toremifene citrate
* Have evidence of prostate cancer (local, regional and/or distal metastasis)
* Have any history of other malignancies (Exceptions include non-melanoma skin cancer or other cancer that has no evidence of tumor reoccurrence 5 years after definitive treatment).
* Have active systemic viral, bacterial, or fungal infections requiring treatment
* Have, in the judgment of the investigator, a clinically significant concurrent illness or psychological, familial, sociological, geographical or other concomitant condition that would not permit adequate follow-up and compliance with the study protocol
* Concurrently being treated with other investigational agents or have participated in an investigational study within 60 days prior to screening
* Currently taking dutasteride. Subject is eligible if he stops dutasteride for a total washout of 90 days prior to the Screening Visit and agrees not to use dutasteride for the duration of the study.
* Have previously taken finasteride for greater than two years
* Currently taking finasteride. Subject is eligible if he stops finasteride for a total washout of 30 days prior to the Screening Visit and agrees not to use finasteride for the duration of the study.
* Currently taking testosterone or testosterone-like supplements, such as dehydroepiandrosterone (DHEA). Subject is eligible if he stops these agents for a total washout of 30 days prior to the Screening Visit and agrees not to use these agents for the duration of the study.
* Have a history of taking PC-SPES within the past two years.
* Currently taking herbal medicine or dietary supplements for prostate health, such as Saw Palmetto (also known as Serenoa Repens).

Subject is eligible if he stops these agents for a total washout of 30 days prior to taking the first dose of study drug and agrees not to use these agents for the duration of the study.

Lycopene, vitamin E and selenium are not prohibited and no washout is required. However, vitamin E intake should be limited to less than 400 i.u. per day.

* Have a history of thromboembolic event or disease including deep vein thrombosis, pulmonary embolus, or thrombotic stroke
* History of chronic hepatitis or cirrhosis

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1589 (Actual)
Dates: Start 2005-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Taneja, MD, Principal Investigator — NYU Langone Medical Center
Locations (138):
- United States (108):
  - Medical Affiliated Research Ctr., Huntsville, Alabama
  - Coastal Clinical Research, Mobile, Alabama
  - Hope Research Inst., Phoenix, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - San Bernardino Urological Associates Medical Group, San Bernardino, California
  - Western Clinical Research, Inc., Torrance, California
  - Urology Research Options, Aurora, Colorado
  - Urology Associates, P.C., Denver, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Connecticut Surgical Group, Hartford, Connecticut
  - Urological Associates of Bridgeport, Trumbull, Connecticut
  - Connecticut Clinical Research, Waterbury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Atlantic Urological Associates, Daytona Beach, Florida
  - Southwest Florida Urologic Associates, Fort Myers, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - UroSearch, Ocala, Florida
  - Central Florida Urology Group/ UroSearch, Ocala, Florida
  - Florida Foundation for Healthcare Research, Ocala, Florida
  - Winter Park Urology Associates, Orlando, Florida
  - Panama City Urological Center, Panama City, Florida
  - Demaur Clinical Research Center, Pembroke Pines, Florida
  - DMI Research, Pinellas Park, Florida
  - Urology Consultants, Pinellas Park, Florida
  - Florida Urology Specialists, Sarasota, Florida
  - Midtown Urology, Atlanta, Georgia
  - Georgia Urology, Atlanta, Georgia
  - Urology Enterprises, Marietta, Georgia
  - North Fulton Urology, Roswell, Georgia
  - St. Joseph's, Candler Health System, Savannah, Georgia
  - Specialty Care Research, Peoria, Illinois
  - Urology of Indiana, LLC, Indianapolis, Indiana
  - Metropolitan Urology, PSC, Jeffersonville, Indiana
  - Kansas City Urology Care, P.C., Overland Park, Kansas
  - Regional Urology, LLC, Shreveport, Louisiana
  - Anne Arundel Urology, Annapolis, Maryland
  - Maryland Prostate Center: University of Maryland Medical Center, Baltimore, Maryland
  - Drs. Werner, Murdock, & Francis PA, Urology Associates, Greenbelt, Maryland
  - Urology Center, PA, Hagerstown, Maryland
  - Mid Atlantic Clinical Research, Rockville, Maryland
  - Chesapeake Urology Research Assoc., Towson, Maryland
  - Brigham & Women's Hospital, Division of Urological Surgery, Boston, Massachusetts
  - Boston Clinical Trials, Brighton, Massachusetts
  - Michigan Medical, PC Urology, Grand Rapids, Michigan
  - Mich. Inst. of Urology, Saint Clair Shores, Michigan
  - Adult & Pediatric Urology, Sartell, Minnesota
  - St. Louis Urological Surgeons, Chesterfield, Missouri
  - Metropolitan Urological Specialists, Florissant, Missouri
  - Midwest Urology Center, Independence, Missouri
  - Washington University Urologic Research Ctr., St Louis, Missouri
  - Urology PC, Lincoln, Nebraska
  - Sheldon Freeman, Las Vegas, Nevada
  - Urologic Surgeons, Ltd., Reno, Nevada
  - Coastal Urology Associates, Brick, New Jersey
  - Central Jersey Clinical Research, Edison, New Jersey
  - Hamilton Urology PA, Hamilton, New Jersey
  - Delaware Valley Urology, Marlton, New Jersey
  - Delaware Valley Urology, Mount Laurel, New Jersey
  - Urology Group of New Mexico, Albuquerque, New Mexico
  - The Urological Institute of Northeastern Research Department, Albany, New York
  - Metropolitan Urologic Services, P.C., Elmont, New York
  - AccuMed Research Associates, Garden City, New York
  - Urological Surgeons of Long Island, Garden City, New York
  - Lake Success Urological Associates, Lake Success, New York
  - Urology Associates, PC, Manhasset, New York
  - NYU Urology Associates, New York, New York
  - University Urology Associates, New York, New York
  - CNY Urology, Oneida, New York
  - Staten Island Urological Research, Staten Island, New York
  - Asheboro Urology Clinic, Asheboro, North Carolina
  - McKay Urology, Charlotte, North Carolina
  - Wake Urology Associates, Raleigh, North Carolina
  - Summa Health System, Cancer Research Office, Akron, Ohio
  - Tri-State Urologic Services/PSC, Inc. d/b/a The Urology Group, Cincinnati, Ohio
  - Capital Urology, Columbus, Ohio
  - Columbus Urology, Inc., Columbus, Ohio
  - Urology of Northern Ohio, Elyria, Ohio
  - Southwest Urology, Middleburg Heights, Ohio
  - Parkhurst Research Organization, Bethany, Oklahoma
  - Urologic Specialists of Oklahoma Research Department, Tulsa, Oklahoma
  - Oregon Urology Specialists, Springfield, Oregon
  - Urologic Associates of Allentown, Allentown, Pennsylvania
  - Urologic Surgery, P.C., Bala-Cynwyd, Pennsylvania
  - Urological Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - The Urology Institute, Monroeville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Triangle Urological Group, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Department of Urology, Pittsburgh, Pennsylvania
  - State College Urologic Associates, Inc., State College, Pennsylvania
  - University Urological Research Institute, Providence, Rhode Island
  - Columbia Urological Associates, Columbia, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Center of the South, Germantown, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Southeast Urology Network, Memphis, Tennessee
  - University of Tennessee, Dept. of Urology, Memphis, Tennessee
  - Urology Associates, Nashville, Tennessee
  - Professional Quality Research, Austin, Texas
  - Research Across America, Dallas, Texas
  - Urology San Antonio Research, PA, San Antonio, Texas
  - Advanced Clinical Research, Salt Lake City, Utah
  - Salt Lake Research, Salt Lake City, Utah
  - Devine-Tidewater Urology, Norfolk, Virginia
  - Med Atlantic, Inc (Virginia Urology), Richmond, Virginia
  - Seattle Urological Associates, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Urologic Northwest Surgeons, Tacoma, Washington
  - Urology Services Madigan Army Medical Center, Tacoma, Washington
- Argentina (6):
  - Centro Urologico Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Pirovano, Buenos Aires
  - Policlinico Bancario de Buenos Aires, Buenos Aires
  - Sanatorio Municipal, Buenos Aires
  - Servicio de Urologia, Buenos Aires
- Canada (24):
  - Prostate Cancer Inst., Calgary, Alberta
  - Alberta Urology Inst.. Research Center, Edmonton, Alberta
  - Southern Interior Medical Research Inc., Kelowna, British Columbia
  - Dr. G. Steinhoff Clinical Research, Victoria, British Columbia
  - Allan B. Patrick, M.D. Professional corporation, Fredericton, New Brunswick
  - Queen Elizabeth Health Sciences Centre, Halifax, Nova Scotia
  - Male/Female Health and Research Centre, Barrie, Ontario
  - Burlington Urology, Burlington, Ontario
  - Centre for Advanced Urological Research, Kingston, Ontario
  - Urology Assoc./Urologic Medical Research, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Mor Urology, Newmarket, Ontario
  - The Fe/Male Health Centres, Oakville, Ontario
  - Urotec, Oshawa, Ontario
  - The Health Institute for Men, Toronto, Ontario
  - Stanley Flax Medical Professional Corp., Toronto, Ontario
  - Univ. Health Network, Princess Margaret Hospital Prostate Centre, Toronto, Ontario
  - The Male Health Centre, Toronto, Ontario
  - Roger Buckley, MD, Willowdale, Ontario
  - Urology South Shore Research, Greenfield Park, Quebec
  - Les Urologues Associes du CHUM, Montreal, Quebec
  - McGill Urology Associates, Montreal, Quebec
  - Ultra-Med, Inc., Pointe-Claire, Quebec
  - G.R.U.M., Trois-Rivières, Quebec

REFERENCES:
- [Derived] Taneja SS, Morton R, Barnette G, Sieber P, Hancock ML, Steiner M. Prostate cancer diagnosis among men with isolated high-grade intraepithelial neoplasia enrolled onto a 3-year prospective phase III clinical trial of oral toremifene. J Clin Oncol. 2013 Feb 10;31(5):523-9. doi: 10.1200/JCO.2012.41.7634. Epub 2013 Jan 7. PMID 23295793

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1,589 subjects were recruited
Groups:
- Placebo: matching placebo
- Toremifene 20mg: toremifene 20mg group tablet q.d.
Period: Overall Study
Arm/Group | Placebo | Toremifene 20mg
Started | 802 | 787
Completed | 598 | 588
Not Completed | 204 | 199
Not completed — Adverse Event | 60 | 64
Not completed — Lost to Follow-up | 23 | 18
Not completed — Physician Decision | 18 | 21
Not completed — Protocol Violation | 13 | 18
Not completed — Withdrawal by Subject | 75 | 70
Not completed — Failure to comply w/dosing regimen | 6 | 4
Not completed — QTc>480 | 3 | 1
Not completed — mililtary deployment | 2 | 0
Not completed — Study Site Closing/PI Moved | 1 | 2
Not completed — Cardiologist recommendation | 1 | 0
Not completed — Pt. moved to another state | 1 | 0
Not completed — Taking exclusionary avodart | 1 | 0
Not completed — Not able to discontinue plavix | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Toremifene 20mg: toremifene 20mg arm
- Placebo: Placebo group
- Total: Total of all reporting groups
Arm/Group | Toremifene 20mg | Placebo | Total
Number analyzed (Participants) | 787 | 802 | 1589
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 425 | 434 | 859
  >=65 years | 362 | 368 | 730
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (7.45) | 64.4 (7.96) | 64.4 (7.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 787 | 802 | 1589
Region of Enrollment [Number; unit: participants]
  United States | 682 | 688 | 1370
  Canada | 97 | 104 | 201
  Argentina | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Toremifene in the Prevention of Prostate Cancer in Men With High Grade Prostatic Intraepithelial Neoplasia (PIN)
Description: To measure the efficacy of toremifene citrate in men with high grade prostatic intraepithelial neoplasia (PIN). Prostate cancer-free survival distributions (Kaplan-Meier)
Time Frame: The outcome measurement time is up to 36 months
Population: MITT: Randomized subjects who were given study drug and did not return it unused and had a baseline and on-study prostate biopsy
Measure: Number (95% Confidence Interval); unit: % of participants cancer-free 36 months
Groups:
- Toremifene 20mg: Toremifene 20mg group
Arm/Group | Placebo | Toremifene 20mg
Number analyzed (Participants) | 717 | 709
% of participants cancer-free 36 months | 54.9 (36.0) [43.3 to 66.5] | 59.5 (36.0) [48.1 to 70.9]

2. Secondary Outcome: The Effect of Toremifene on Lipid Levels
Description: Measure lipid levels including total cholesterol, LDL, HDL and Triglycerides % change from baseline
Time Frame: Up to 36 months
Population: All randomized subjects who take at least 1 dose of study drug
Measure: Mean (Standard Deviation); unit: % of change
Arm/Group | Placebo | Toremifene 20mg
Number analyzed (Participants) | 802 | 787
% of change
  Cholesterol | -3.678 (18.2317) | -6.675 (116.9705)
  LDL | -7.447 (64.8765) | -7.824 (28.8209)
  HDL | 3.69 (19.133) | 0.29 (16.650)
  Triglycerides | 16.298 (58.003) | 0.319 (47.9793)

3. Secondary Outcome: The Effect of Toremifene on Hormone Levels
Description: % Change from baseline hormone levels, including total testosterone, free testosterone, dihydrotestosterone (DHT) and estradiol
Time Frame: Up to 36 months
Population: Any randomized subject taking at least 1 dose of study drug
Measure: Mean (Standard Deviation); unit: % of change
Arm/Group | Placebo | Toremifene 20mg
Number analyzed (Participants) | 802 | 787
% of change
  DHT | 17.736 (48.3284) | 46.409 (60.2061)
  Estradiol | 11.9 (67.86) | 53.2 (151.5)
  Testosterone total | 2.246 (102.9086) | 31.136 (63.5961)
  Testosterone free | 17.71 (438.652) | 7.92 (65.114)

4. Secondary Outcome: The Effect of Toremifene on Total PSA (Prostate Specific Antigen) Levels
Description: To assess the effect of toremifene in the total PSA (prostate specific antigen) levels from baseline
Time Frame: Up to 36 months
Population: Any randomized subject taking at least 1 dose of study drug
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Placebo | Toremifene 20mg
Number analyzed (Participants) | 790 | 776
mcg/L | 0.82 (7.360) | 1.07 (3.632)

5. Secondary Outcome: The Effect of Toremifene on the Mean Change at 36 Months in AUA (American Urological Association) Symptom Score
Description: To assess the effect of toremifene on the AUA (American Urological Association) symptom score mean change from baseline. Scores of 0-7=mild severity, 8-9, moderate, and 20-30, severe with possible responses of 0 (not at all) 1 (<1/5), 2 (<50% time), 3 (about 50% time), 4 (> 50% time) & 5 (Almost Always). There are 7 questions (1)Incomplete emptying (2)Frequency (3)Intermittency (4)Urgency (5)Weak-stream (6)Straining & (7)Nocturia. Analysis is change from baseline at final evaluation (36 months) for quality of life due to urinary symptoms. The P Value is from a Wilcoxon signed-rank test. Scores can range from 0-35, highest representing worse symptoms
Time Frame: 36 months
Population: Reference to J Urol.1992 Nov;148(5):1549-57; discussion 1564. AUA symptom index for benign prostatic hyperplasia. The Measurement Committee of the American Urological Assocciation.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Toremifene 20mg
Number analyzed (Participants) | 676 | 653
scores on a scale | 1.1 (5.4) | 1.2 (5.6)

6. Primary Outcome: Occurrence of a Positive Cancer Biopsy
Description: To measure the occurrence of a positive cancer biopsy
Time Frame: Up to 36 months
Population: Modified, intend-to-treat (MITT) all randomized subj. who take at least 1 dose of study drug, and had baseline and on-study prostate biopsies, where the baseline biopsy did not have cancer.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Placebo: Determine occurrence of positive cancer biopsy
- 20 mg. Toremifene: Determine occurrence of positive cancer biopsy and survival time
Arm/Group | Placebo | 20 mg. Toremifene
Number analyzed (Participants) | 717 | 709
Months | 23.5 [8.8 to 32] | 15.9 [11.1 to 33]

7. Secondary Outcome: Occurrence of High Grade PIN at the 12, 24, 36 Month Biopsies
Description: To measure the occurrence of high grade PIN at the 12, 24, 36 Month intervals in the 360 days study.
Time Frame: Up to 36 months
Population: All randomized subjects that took 1 dose of study drug
Measure: Number; unit: Subjects
Arm/Group | Placebo | Toremifene 20mg
Number analyzed (Participants) | 802 | 787
Subjects
  12 months | 167 | 149
  24 months | 90 | 103
  36 months | 92 | 94

8. Secondary Outcome: The Effect of Toremifene on % Free Serum PSA (Prostate Specific Antigen) Levels, Change From Baseline
Description: To assess the effect of toremifene in % free serum PSA (prostate specific antigen) levels, change from baseline
Time Frame: 36 months
Population: Any randomized subject taking at least 1 dose of study drug
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Placebo | Toremifene 20mg
Number analyzed (Participants) | 358 | 356
mcg/L | 2.3 (11.24) | 2.0 (10.49)

ADVERSE EVENTS:
Time Frame: Three years
Arm/Group | Placebo | Toremifene 20mg
Serious Adverse Events (participants affected / at risk) | 137/802 | 117/787
Other Adverse Events (participants affected / at risk) | 666/802 | 631/787
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=802) | Toremifene 20mg (N=787)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina Pectoris (Endocrine disorders) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 2 (2)
Aortic Valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 4 (4) | 5 (5)
Atrial Flutter (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac Disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 2 (3) | 2 (3)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 15 (16) | 7 (7)
Hypertrophic obstructive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 6 (6) | 2 (2)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Idiopathic Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis perforated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 5 (5) | 3 (3)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2)
Bronchititis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Central line infection (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 1 (1)
Clostridium colitis (Infections and infestations) | 1 (1) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Human ehrlichiosis (Infections and infestations) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 6 (7)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0)
Postoperative infection (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 4 (4)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Urosepsis (Infections and infestations) | 4 (4) | 6 (6)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Device failure (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nerve root injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Surgical procedure repeated (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus insulin-dependent (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (5)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (11) | 6 (6)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell carcinoma of the kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 2 (2)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 2 (2)
Major depression (Psychiatric disorders) | 0 (0) | 1 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder diverticulum (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 3 (3)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=802) | Toremifene 20mg (N=787)
Hypertension (Vascular disorders) | 70 (70) | 52 (52)
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 (61) | 46 (50)
Urinary tract infection (Infections and infestations) | 54 (65) | 41 (45)
Upper respiratory tract infection (Infections and infestations) | 46 (57) | 45 (53)
Prostatitis (Reproductive system and breast disorders) | 49 (62) | 39 (43)
Erectile dysfunction (Reproductive system and breast disorders) | 42 (42) | 42 (43)
Haematuria (Renal and urinary disorders) | 38 (49) | 36 (43)
Back pain (Musculoskeletal and connective tissue disorders) | 36 (41) | 31 (32)
Dizziness (Nervous system disorders) | 37 (42) | 30 (32)
Nasopharyngitis (Infections and infestations) | 39 (42) | 28 (30)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 30 (31) | 32 (32)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 (29) | 32 (34)
Fatigue (General disorders) | 31 (32) | 28 (28)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 32 (34) | 24 (24)
Pollakiuria (Renal and urinary disorders) | 30 (30) | 26 (27)
Cataract (Eye disorders) | 24 (32) | 29 (37)
Insomnia (Psychiatric disorders) | 32 (34) | 21 (21)
Sinusitis (Infections and infestations) | 21 (23) | 32 (34)
Urinary retention (Renal and urinary disorders) | 24 (28) | 29 (34)
Constipation (Gastrointestinal disorders) | 27 (27) | 24 (24)
Headache (Nervous system disorders) | 27 (29) | 22 (27)
Nocturia (Renal and urinary disorders) | 23 (24) | 25 (26)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 26 (26) | 21 (21)
Nausea (Gastrointestinal disorders) | 26 (29) | 21 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction: PIs may publish/present trial results at med. conferences after 1st of 1 of following occurs: complete Multicenter Study publication presented/Sponsor confirms there won't be Multicenter Study publication/18 mos. elapsed after Study ends. PI:submits advance copy w/in 60 days. Sponsor:60 days to review. Sponsor:tells PI w/in 60 days the pres./pub. might have adverse effect to obtain patents on inventions or confidentiality of info, PI can't make pres/pub w/o changes